CLINICAL TRIAL: NCT05554679
Title: Maternal and Fetal Outcome With Metformin Therapy for Obese Pregnant Women a Randomized Control Trial.
Brief Title: Maternal and Fetal Outcome With Metformin Therapy for Obese Pregnant Women .
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: financial issues
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Ibram Samy, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Metformin in preganancy
Record Dates: First submitted 2020-03-20; First posted 2022-09-26 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Metformin for Obese Pregnant Women
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Intervention Model Description: metformin effect on prevention of macrosomia in obese pregnant women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): obese pregnant women who take metformin
  Interventions: Drug: Metformin
- group B (No Intervention): obese pregnant women who take no metformin

INTERVENTIONS:
Drug: Metformin — Metformin is an oral insulin-sensitising medication that acts to decrease blood glucose concentrations. It inhibits pathways in the liver that stimulate glucose production and also acts to increase glucose uptake into skeletal muscle and fat cells . Metformin is commonly used in the treatment of type 2 diabetes mellitus and polycystic ovarian syndrome , and is being used increasingly in the treatment of gestational diabetes, having been shown to result in decreased rates of neonatal hypoglycaemia and no increased risk of adverse maternal outcomes when compared with insulin.
  Arms: group A

SUMMARY:
To evaluate the role of metformin in pregnant women with obesity (BMI above 30) , on maternal and infant outcome.

DETAILED DESCRIPTION:
Obesity is defined as having an excessive amount of body fat based on the BMI, Obesity can be classified based on the BMI to obese class I ,Class II ,and extreme obesity (class III) , Obesity can harm the fertility by inhibiting normal ovulation. Even in women who regularly ovulate, the greater the BMI, the longer it appears to take to become pregnant. Obesity can also affect the outcome of in vitro fertilization (IVF). (1)

Being obese during pregnancy increases the risk of various pregnancy complications, including :

Miscarriage ,stillbirth ,GD , preeclampsia , obstructive sleep apnea , difficult vaginal delivery ,need for C-section ,and complication of C-section ,Fetal macrosomia , and increasing the risk for metabolic syndrome and childhood obesity , it also make It may be hard for the participants health care provider to diagnose birth defects during pregnancy even prenatal tests like ultrasound(2),(3) .

Normal weight gain during pregnancy for obese women having single pregnancy is between about (5-9) KG .

Normal weight gain during pregnancy for obese women having Multiple pregnancy is between about (11-19) KG (4).

For women who are extremely obese, gaining less than the recommended amount or losing weight during pregnancy might lower the risk of fetal and neonatal macrosomia .

The fetus is regarded as suspected appropriate or gestational age (AGA) when the Sonographic Estimated Fetal Weight (SEFW) is at 10th to 90th percentile for gestational age (GA), and suspected LGA when the SEFW > 90th percentile (5) .

A baby diagnosed with fetal macrosomia has a birth weight of more than 8 pounds,(4,000 grams), regardless of his or her gestational age (6,7,8) .

In this study the investigator will try to focus on diagnose undiagnosed diabetic using GTT (glucose tolerance test specially with women who has one or more risk factors A raised body mass index (BMI) over 30kg/m². A previous baby over 4kg or more ,Confirmed gestational diabetes in a previous pregnancy or have a first degree relative that has diabetes All pregnant women who have not already been diagnosed with diabetes should be screened for Diabetes with a fasting plasma glucose (FPG), an HbA1c, or an untimed random plasma glucose test at their first prenatal visit

* Women who by 24 weeks' gestation have not yet been diagnosed with overt or gestational diabetes should, at between 24 and 28 weeks' gestation, undergo a 2-hour, 75-g OGTT for gestational diabetes
* At 24-28 weeks' gestation, a result of 153-199 mg/dL for a 2-hour, 75-g OGTT indicates gestational diabetes, while a test result of 200 mg/dL or higher indicates overt diabetes(9),(10)

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with BMI ≥ 30 kg/m2, and normal glucose tolerance test.

Exclusion Criteria:

* pregnant women who are diabetic,
* had a history of previous GDM,
* previous small baby,
* PCO or
* previous early pre-eclampsia,

Ages: 17 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 178 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Neonatal birth weight | Baseline
  The fetus is regarded as suspected appropriate for gestational age (AGA) when the Sonographic Estimated Fetal Weight (SEFW) is at 10th to 90th percentile for gestational age (GA), and suspected LGA when the SEFW > 90th percentile ,A baby diagnosed with fetal macrosomia has a birth weight of more than 8 pounds,(4,000 grams), regardless of his or her gestational age.

SECONDARY OUTCOMES:
Maternal weight gain | Baseline
  Health care providers who care for pregnant women should determine a woman's body mass index at the initial prenatal visit and counsel her regarding the benefits of appropriate weight gain, nutrition and exercise, and, especially, the need to limit excessive weight gain to achieve best pregnancy outcome . for women of normal weight, 14.1-22.7 kg (31-50 lb) for overweight women, and 11.3-19.1 kg (25-42 lb) for obese women

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abuelhasan, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Hyer S, Balani J, Shehata H. Metformin in Pregnancy: Mechanisms and Clinical Applications. Int J Mol Sci. 2018 Jul 4;19(7):1954. doi: 10.3390/ijms19071954. PMID 29973490